

## QUALITY OF LIFE AND PSYCHOLOGICAL STRENGTHS OF OLDER PEOPLE: ASSESSMENT AND INTERVENTION



## PATIENT INFORMTION DOCUMENT AND INFORMED CONSENT

**Research project:** "QUALITY OF LIFE AND PSYCHOLOGICAL STRENGTHS OF THE ELDERLY. EVALUATION AND INTERVENTION".

## 1) Information to the patient about the object of the study:

The study is being carried out by professors of the Department of Psychology of the CEU San Pablo University of Madrid. Its main purpose is to focus on the psychological strengths of people to cope with stressful situations.

To this end, some components such as quality of life, psychological well-being, emotional distress, acceptance, resilience, gratitude, the way in which situations are faced, as well as sociodemographic variables, health and family functioning and loneliness are analyzed. The benefits of these results will allow us to know the protective or risk factors with which to develop prevention and intervention programs with different age groups. The study does not imply any risk for the participants, their participation is completely voluntary.

Your participation in the study will consist of answering the following questions in a questionnaire created to evaluate the aspects mentioned above. This is a short questionnaire that lasts approximately 30 minutes.

At the end of the questionnaire you will be asked a question "Would you be interested in continuing to collaborate in this investigation?

- a. If the answer is negative, i.e., you do not want to continue collaborating, your participation ends here and this data would be anonymous, since we would have no way of identifying the person.
- b. If the answer is affirmative, that is, you want to continue collaborating, we need you to provide us with your e-mail address or telephone number so that we can send you the questionnaire again in which your participation will be required. In this case the data will be pseudonymized. This means that the column in which your email or telephone number appears will be removed from that database and copied to another Excel database that will be encrypted and a random code will be assigned to each participant who has provided their contact information. Therefore, the information will be processed without being able to identify any participant at any time.



When contacting the participants who agreed to continue collaborating, the encrypted document will be accessed again to access this information and proceed with the next step.

## 2) Informed consent:

- 1. I have read and understood the information sheet that is the subject of the study.
- 2. I have had the opportunity to ask questions.
- 3. My questions have been answered to my satisfaction.
- 4. I have received sufficient information about the study and the tests to be performed.
- 5. I understand that participation is voluntary and I can leave the study whenever I wish without having to give explanations and without affecting my medical care.
- 6. In accordance with the provisions of Regulation (EU) 2016/679 of the European Parliament and of the Council of 27 April 2016 on the protection of natural persons with regard to the processing of personal data and on the free movement of such data and repealing Directive 95/46/EC, as well as other current and applicable regulations on the protection of personal data, I have been informed that my personal data, obtained through the completion of this form as well as those resulting from my participation in the project will be processed under the responsibility of the FUNDACIÓN UNIVERSITARIA SAN PABLO CEU (hereinafter, FUSP-CEU), in order to manage my participation in this research project.

In addition, I have been informed of the following aspects:

- a. That the elaboration of profiles is foreseen in order to analyze or predict aspects related to my health.
- b. That the treatments indicated are legitimized by the consent given by me.
- c. That my personal data, obtained by filling in this form, as well as those resulting from my participation in the project will be kept for the time necessary for the development of this research, which is estimated to be 12 months, and will be subsequently destroyed, without being able to be kept without having been previously anonymized. In any case, they cannot be transferred without my express consent and I do not give it in this act.



- d. That I can contact the Data Protection Delegate of FUSP-CEU, by sending my request in writing to the postal address C/ Tutor no 35 -28008 Madrid or to the e-mail address dpd@ceu.es.
- e. That in accordance with the rights conferred on me by current data protection regulations, I may contact the competent Control Authority to file the claim I deem appropriate, as well as exercise my rights of access, rectification, limitation of processing, deletion, portability and opposition to the processing of my personal data and withdraw the consent given for the processing of the same, by sending my request to the researcher responsible at the contact address given in this document.
- 7. I agree that my written consent and other data will be available to the clinical research project in which I am participating, and to the researchers responsible for it, Gema Pérez Rojo and Javier López Martínez, but always respecting confidentiality and the guarantee that my data will not be publicly available so that I can be identified.
- 8. The data collected for this study will be included, with those of other persons participating in this study, in a personal database of the CEU University, to which only the researchers approved for this project will have access, all of them being subject to the secrecy inherent to their profession or derived from a confidentiality agreement.
- 9. I sign this information and consent document voluntarily to express my desire to participate in this research study until I decide otherwise. By signing this consent, I do not waive any of my rights and I will receive a copy of this document for future reference.

| Patient's name and surname: | |
|------------------------------------------|-----------------------|
| ID card/Passport: | |
| Signature: | <u>Date</u> : |
| Name and surname of the legal representa | ative, if applicable: |
| ID card/Passport: | |
| Signature: | Date: |



Name and surname of the researcher: Javier López Martínez

ID card: 16301728H

Researcher's contact address: Universidad CEU San Pablo, Campus de Montepríncipe (Alcorcón) Facultad de Medicina, Departamento de Psicología y Pedagogía, Despacho 0029 Pabellón MED.

E-mail: jlopezm@ceu.es

Name and surname of the researcher: Gema Pérez Rojo DNI 53046948R

Researcher's contact address: Universidad CEU San Pablo, Campus deMontepríncipe (Alcorcón) Facultad de Medicina, Departamento de Psicología y Pedagogía, Despacho 0029 Pabellón MED.

E-mail: gema.perezrojo@ceu.es

V° B° of the Study Director (or Principal Investigator of the study):